CLINICAL TRIAL: NCT07269782
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX43 (Anti-PD-L1 ADC) in Combination With Serplulimab as Neoadjuvant Therapy in Subjects With NSCLC
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of HLX43 + Serplulimab as Neoadjuvant Therapy in Subjects With NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-NSCLC203
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX43 DOSE 1 + Serplulimab (Experimental): Patients will receive the treatment once every 3 weeks (Q3W), for 4 cycles.
  Interventions: Drug: HLX43 DOSE 1; Drug: Serplulimab
- HLX43 DOSE 2 + Serplulimab (Experimental): Patients will receive the treatment once every 3 weeks (Q3W), for 4 cycles.
  Interventions: Drug: HLX43 DOSE 2; Drug: Serplulimab

INTERVENTIONS:
Drug: HLX43 DOSE 1 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Anti-PD-L1 ADC
  Arms: HLX43 DOSE 1 + Serplulimab
Drug: HLX43 DOSE 2 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Anti-PD-L1 ADC
  Arms: HLX43 DOSE 2 + Serplulimab
Drug: Serplulimab — Serplulimab Injection, Recombinant humanized anti PD 1 monoclonal antibody
  Other Names: HLX10

SUMMARY:
The study is being conducted to to explore the reasonable dosage and evaluate the efficacy and safety of HLX43 (Anti-PD-L1 ADC) in Combination with Serplulimab (Anti-PD-1 Recombinant Humanized Monoclonal Antibody) as Neoadjuvant Therapy in Subjects with Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
This study is a randomized, open-label phase II clinical study to explore the reasonable dosage and evaluate the efficacy and safety of HLX43 (Anti-PD-L1 ADC) in Combination with Serplulimab (Anti-PD-1 Recombinant Humanized Monoclonal Antibody) as Neoadjuvant Therapy in Subjects with Non-Small Cell Lung Cancer (NSCLC)，In this study, eligible subjects will be randomized at 1:1 ratio, and the patients will be administered with HLX43 at one of the two dose levels plus Serplulimab at a fixed dosage via intravenous infusion every 3 weeks (Q3W) for 4 cycle.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a full understanding of the study content, process, and possible adverse reactions before the study, and sign the informed consent form (ICF); voluntarily participate in the study; be able to complete the study as per protocol requirements;
* 2. Aged ≥ 18 years and ≤ 75 years at the time of signing the ICF, male or female;
* 3. Histologically or cytologically confirmed NSCLC;
* 4. Diagnosed with stage II-IIIB NSCLC (according to the Union for International Cancer Control and the American Joint Committee on Cancer (AJCC) TNM staging system for lung cancer (8th edition)), without actionable genomic alterations (AGAs); subjects with non-squamous NSCLC must have previous test results confirming negative EGFR and ALK gene alterations, and if no previous EGFR and ALK test results are available, the subjects are required to undergo relevant tests at the study site; for subjects with squamous NSCLC, if the previous EGFR and/or ALK gene status is unknown, corresponding tests are not required before enrollment in this study;
* 5. Agree to undergo surgery if eligible after neoadjuvant therapy; prior to study enrollment, the subject should be assessed by the primary thoracic surgeon, who holds the main responsibility for the surgery, to confirm eligibility for R0 resection with curative intent as required by the study; the subject must have good cardiac function and be confirmed as eligible for surgical resection with curative intent;
* 6. At least one measurable lesion as per RECIST 1.1 within 4 weeks prior to randomization;
* 7. Subjects who agree to provide archived tumor tissue specimens that meet the testing requirements (either from the most recent surgery or biopsy, preferably within 2 years) or agree to undergo a biopsy to collect tumor tissue for PD-L1 expression testing; Note: Formalin-fixed paraffin-embedded (FFPE) tumor samples (paraffin blocks or unstained sections, which must meet the quality control criteria for testing) from the most recent surgery or biopsy at or after the diagnosis of malignant tumor and pathological reports of such specimens should be provided by subjects.
* 8. The following conditions must be met in terms of the time of the first administration of the investigational product: at least 3 weeks from the previous major surgery or medical device treatment; at least 1 week from the previous minor surgery; recovery of treatment-induced AEs to Grade ≤ 1 (CTCAE v5.0);
* 9. ECOG PS score of 0-1 within one week prior to randomization;
* 10. Life expectancy > 3 months;
* 11. Adequate organ functions as confirmed by laboratory tests within 1 week prior to randomization (no blood transfusions or treatment with albumin, recombinant human thrombopoietin, or colony-stimulating factor (CSF) within 14 days prior to the first dose)；
* 12. Male and female subjects with childbearing potential must agree to use at least one highly effective contraception method during the study and within at least 6 months after the last dose of the investigational product; female subjects of childbearing age must be negative for pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* 1. Histologically or cytologically confirmed tumor containing components of small cell lung cancer or neuroendocrine carcinoma;
* 2. Any prior systemic or local anti-tumor therapy for non-small cell lung cancer, including chemotherapy, radiotherapy, or immunotherapy;
* 3. History of any second malignancy within 2 years prior to randomization, except for early-stage malignancies (carcinoma in situ or stage I tumors) that have received radical treatment, such as non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma;
* 4. History of adverse events leading to permanent discontinuation of immunotherapy, or history of ≥ Grade 2 immune-related pneumonitis or immune-related myocarditis;
* 5. Subjects with current or prior history of clinically significant pulmonary impairment due to pulmonary comorbidities, including but not limited to any underlying lung disease (e.g., pulmonary embolism within 3 months prior to the first dose, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, interstitial pneumonitis, pneumoconiosis, drug-related pneumonitis, and pleural effusion), any autoimmune, connective tissue, or inflammatory disease that may involve the lungs (i.e., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis), prior pneumonectomy that may interfere with the detection and management of suspected drug-related pulmonary toxicity, or history of radiation pneumonitis within 6 months;
* 6. Patients with any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (1) NYHA Class II or greater heart failure or left ventricular ejection fraction (LVEF) < 50%; (2) unstable angina pectoris; (3) myocardial infarction or cerebrovascular accident within 6 months (except lacunar infarction, slight cerebral ischemia, or transient ischemic attack); (4) poorly controlled arrhythmia (including QTc interval ≥ 470 ms) (QTc interval is calculated by Fridericia's formula); (5) poorly-controlled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg after active treatment);
* 7. Patients with active systemic infectious diseases requiring intravenous antibiotics within 2 weeks prior to randomization;
* 8. Patients who have previously received other antibodies/drugs against immune checkpoints, such as PD-1, PD-L1, CTLA4, etc.;
* 9. Patients who have used moderate or potent CYP2D6 or CYP3A inhibitors or inducers within 2 weeks prior to randomization;
* 10. Patients who have received systemic corticosteroids (prednisone > 10 mg/d or equivalent dose of similar drug) or other immunosuppressants within 2 weeks prior to randomization; Except: patients treated with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; short-term prophylactic use of corticosteroids for contrast agents, etc.;
* 11. Patients with known active or suspected autoimmune diseases. Patients with autoimmune-related hypothyroidism and receiving thyroid hormone replacement therapy and those with type 1 diabetes mellitus controlled with insulin therapy are eligible to be enrolled;
* 12. Patients who have received a live vaccine or live attenuated vaccine within 4 weeks prior to randomization;
* 13. Patients who are known to have anaphylaxis to macromolecular protein preparations/monoclonal antibodies or are allergic to any component in the formulation of the investigational product;
* 14. Patients with active tuberculosis;
* 15. Patients with a history of immunodeficiency, including human immunodeficiency virus (HIV)-positive or other acquired or congenital immunodeficiencies, or history of organ transplantation;
* 16. Patients with active HBV or HCV infection or HBV/HCV co-infection; Note: Patients who test positive for HBsAg or HBcAb during the screening period must undergo further HBV-DNA testing, and may be enrolled only if the test result indicates < 500 IU/mL, < 2500 copies/mL, or < ULN. Patients with detectable HBV-DNA must agree to receive treatment with anti-HBV nucleos(t)ide analogs during the study.

Patients who test positive for HCV antibody must undergo further HCV-RNA testing, and may be enrolled only if the test result indicates < ULN.

Patients with HBV/HCV co-infection (positive test for HBsAg or HBcAb and positive test for HCV antibody) should be excluded.

* 17. Pregnant or lactating women;
* 18. Patients who are not suitable for participating in this clinical study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
MPR | At time of surgery
  The percentage of residual viable tumor cells ≤ 10% in the resected primary lesion after neoadjuvant therapy, regardless of the presence of residual viable tumor cells in the lymph nodes.

SECONDARY OUTCOMES:
PCR | At time of surgery
  The absence of residual viable tumor cells in both the resected primary lesion and lymph nodes after neoadjuvant therapy.
ORR | up to 12 week
  Objective response rate (ORR) is the proportion of subjects with the best overall response being CR or PR (assessed by investigator per RECIST v1.1)
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, Dr, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China